CLINICAL TRIAL: NCT00435149
Title: Post-operative Mobilization for Carpal Tunnel
Brief Title: Post-operative Mobilization for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Dr. Donald Lee, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 060974
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Carpal tunnel release surgery
- 2 (Active Comparator)
  Interventions: Procedure: Carpal tunnel release surgery

INTERVENTIONS:
Procedure: Carpal tunnel release surgery — Patient will have carpal tunnel release surgery and will be put in a splint after surgery.
  Arms: 1
Procedure: Carpal tunnel release surgery — Patient will have carpal tunnel release surgery and will have a bandage placed over the incision site after surgery.
  Arms: 2

SUMMARY:
This study will investigate the effect of one week of immobilization following carpal tunnel release surgery versus no immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open carpal tunnel release will be included in this study.
* Patients must have clinical evidence of carpal tunnel syndrome.
* Patients must have positive EMG results.
* English speaking patients only.

Patient selection factors include:

* Ability and willingness to follow instructions.
* Patients who are able and willing to return for follow-up evaluations.
* Patients of all races and genders.
* Patients who are able to follow care instructions.

Exclusion Criteria:

* Patients less than 18 years old.
* Patients who are pregnant.
* Patients unwilling or unable to comply with a rehabilitation program for carpal tunnel release who indicate difficulty or inability to return for follow-up visits prescribed by the study protocol.
* Patients who qualify for inclusion in the study, but refuse consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Function assessment questionnaire score, pain score questionnaire, and measurements will be used to determine outcome. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie Daniels, BBA, Study Director — VUMC
Locations (1):
- Vanderbilt Orthopaedic Institute, Nashville, Tennessee, United States